CLINICAL TRIAL: NCT06896461
Title: Validation of Lung Surfactant Protein Type B Levels As a Diagnostic and Prognostic Marker in Heart Failure Progression
Brief Title: Surfactant Derived Protocol in Heart Failure
Acronym: (SPB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Ospedale San Luca, Istituto Auxologico Italiano, Milano (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCM470
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Exercise Test; Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Heart failure patients (Experimental): All heart failure patients wll be charachterized according to cardiopulmonary exercise test variables, spirometry and biomarkers collection
  Interventions: Diagnostic Test: Cardiopulmonary exercise test; Diagnostic Test: Lung function; Diagnostic Test: Biomarkers evaluation

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test — The test consists of physical exertion performed on a stationary bike with a progressively increasing workload, continuing until specific electrocardiographic and/or clinical criteria are met or muscle fatigue occurs. The rate of workload increase (ramp) will be personalized and adjusted to ensure the exercise reaches its peak in approximately 10 minutes.
  Throughout the test, a continuous electrocardiogram (ECG) will be recorded, and various physiological parameters will be measured. These include ventilation, oxygen consumption, carbon dioxide production, and related derived parameters, which will be assessed using a mouthpiece or a face mask through which you will need to breathe for the entire duration of the test. Blood pressure will also be measured at two-minute intervals.
Diagnostic Test: Lung function — Assessment of both static lung volumes (vital capacity, total lung capacity, functional residual capacity, and residual volume) and dynamic lung volumes (forced vital capacity and forced expiratory volume in one second, or FEV1).
  Additionally, the flow-volume curve is measured, generated by continuously recording airflow and volume using an electronic spirometer during a foThe diffusion capacity for carbon monoxide (DLCO) can be measured using the single-breath method (DLCOSB). The patient inhales a small, known concentration of carbon monoxide (CO), holds their breath for 10 seconds, and then exhales. A sample of alveolar gas (from the end of expiration) is analyzed to determine the amount of CO absorbed during the breath, expressed in ml/min/mm Hg.
  By repeating the test with inhalation of gas mixtures containing different oxygen concentrations (approximately 20%, 40%, and 60%), it is possible to assess the diffusion subcomponents: the membrane component and capillary blood volume.
Diagnostic Test: Biomarkers evaluation — Samples of plasma will be collected for bimarkers quantification in heart failure.
  Speecifically, plasma levels will be quantitatively assessed using plasma obtained from venous blood. Blood will be collected in tubes containing 0.129 M Na-citrate (9 volumes of blood to 1 volume of Na-citrate), immediately centrifuged at 3000 g for 15 minutes at 4°C. Circulating levels of both immature and mature SP-B will be analyzed via Tricine gel electrophoresis followed by immunoblotting with an anti-SP-B antibody, allowing for the detection of all SP-B isoforms (proprotein 42 kDa, intermediate 23 kDa, and mature 8 kDa).
  To validate potential heart failure biomarkers, a quantitative, scalable, and cost-effective method-Multiple Reaction Monitoring (MRM)-will be used. MRM, based on triple quadrupole mass spectrometry, enables precise quantification of proteins/peptides and their isoforms in complex biological samples.

SUMMARY:
Pulmonary surfactant is a highly surface-active lipoprotein complex that lines the alveoli and terminal airways, reducing surface tension and preventing alveolar collapse at the end of expiration. It consists of a lipid (90%) and a protein fraction, with surfactant proteins SP-A, SP-B, SP-C, and SP-D playing crucial roles. SP-B is essential for surfactant function, and its absence leads to severe respiratory failure. Recent studies have shown that plasma SP-B levels are elevated in heart failure (HF) patients, likely due to increased pulmonary microvascular pressure and alveolar-capillary barrier dysfunction. SP-B correlates with HF severity and prognosis, outperforming functional parameters as a predictor of hospitalization. This study aims to compare surfactant proteins with other biomarkers, including RAGE, a receptor linked to lung injury. Using advanced multiplex mass spectrometry, the study seeks to validate immature SP-B as a reliable diagnostic and prognostic marker for HF.

DETAILED DESCRIPTION:
Pulmonary surfactant is a highly surface-active lipoprotein complex that forms a thin film lining the alveolar and terminal airway surfaces. Its primary physiological function is to reduce surface tension at the air-liquid interface, stabilizing the alveoli and preventing their collapse at the end of expiration. Both the lipid and protein fractions of surfactant are synthesized by type II pneumocytes and stored in lamellar bodies-intracellular organelles where surfactant is secreted through the fusion of their outer membrane with the apical plasma membrane of the cell, releasing surfactant into the alveolar space.

The surface-active properties of pulmonary surfactant at the liquid-gas interface of the alveoli are primarily attributed to its lipid component (90%), particularly phospholipids. Although accounting for less than 10% of the surfactant, the protein fraction-composed of SP-A, SP-B, SP-C, and SP-D-plays a crucial role. SP-B, along with SP-C, is essential for the lipid fraction's ability to exert its surface-active function. The absence of SP-B is associated with severe respiratory failure, which can be fatal. SP-A and SP-D are less directly involved in surfactant's surface activity but appear to have significant anti-infective functions in the lungs.

Human SP-B is a small amphipathic peptide of 79 amino acids (8 kDa), produced through proteolytic processing from a 381-amino acid precursor (42 kDa). It is encoded by a single gene (SFTPB) located on chromosome 2. SP-B is predominantly produced by type II alveolar epithelial cells, initially synthesized as a glycosylated precursor that is transported from the endoplasmic reticulum to the Golgi apparatus, then to multivesicular bodies, and finally packaged into lamellar bodies. The proteolytic maturation of SP-B occurs during its transfer from multivesicular bodies to lamellar bodies, where active SP-B is stored together with SP-C and phospholipids. The contents of lamellar bodies are secreted into the airway space, where SP-A facilitates surfactant film formation over the alveolar surface.

Extracellular SP-B plays a fundamental role in surfactant homeostasis by promoting lipid absorption into the surface film and enhancing its stability during the compression and expansion cycles of respiration.

Recent studies have shown that in heart failure (HF) patients, plasma SP-B levels are significantly elevated, likely due to increased pulmonary microvascular pressure, which may compromise alveolar-capillary barrier integrity, leading to SP-B release into circulation. Plasma levels of immature SP-B, a surfactant protein isoform, increase in HF patients and strongly correlate with functional indicators of pulmonary impairment (peak oxygen uptake, VO2, lung diffusion, DLco) and New York Heart Association (NYHA) classification, establishing SP-B as a specific marker of disease severity linked to organ damage. More importantly, our studies indicate that SP-B is a circulating prognostic marker for hospitalization in HF patients, with superior predictive ability compared to functional parameters. Furthermore, SP-B also emerges as a marker of therapeutic efficacy.

Despite extensive research, the availability of diagnostic biomarkers for HF remains limited. In addition to natriuretic peptides, which vary under different pathological conditions and lack specificity for HF, a limited number of novel biomarkers have recently emerged, including interleukine ST2, Growth/differentiation factor 15 (GDF-15), Cystatin C, lipocalina-2 (NGAL), and Galectin-3.

Additionally, circulating levels of surfactant protein D (SP-D), which typically increase in pulmonary inflammation, asthma, emphysema, or chronic obstructive pulmonary disease (COPD), have been linked to cardiovascular disease and overall mortality in patients with coronary artery disease diagnosed via angiography. These associations appear independent of conventional risk factors such as age, smoking, cholesterol levels, and C-reactive protein.

This study aims to compare surfactant protein levels with previously described biomarkers and with RAGE (Receptor for Advanced Glycation End Products), a surface molecule belonging to the immunoglobulin superfamily. Unlike other receptors, RAGE is characterized by its multi-ligand nature, allowing interactions with various molecules involved in homeostasis, development, and inflammation. Recent findings indicate that RAGE levels are altered in pulmonary damage conditions such as sarcoidosis, pulmonary fibrosis, and chronic bronchitis, suggesting its potential role as an organ damage marker.

By employing advanced multiplexing methodology based on mass spectrometry, this study will validate the role of immature SP-B as a precise diagnostic and prognostic biomarker for heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure diagnosis
* Left ventricular ejection fraction <40%
* Stable clinical condition

Exclusion Criteria:

* Relevant comorbidities
* usual contraindications to cardiopulmonary testing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of lung surfactant protein type B levels in heart failure by multiplexing methodology | 2 years
  analyses will be carried out using modern multiplexing methodology based on mass spectrometry, that will make it possible to validate the role of the immature SP-B protein as an accurate marker for the diagnosis and prognosis of heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided